CLINICAL TRIAL: NCT02145598
Title: Phase II Study of Bortezomib, Melphalan, Prednisone (VMP) Followed by Lenalidomide Maintenance vs. VMP Without Maintenance in Myeloma Patients Not Eligible to High-dose Chemotherapy and Autologous Stem Cell Transplantation
Brief Title: Treatment Optimization in Patients With Untreated Multiple Myeloma
Acronym: GERMAIN
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Dr. med. Lars-Olof Muegge (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Lars-Olof Muegge, MD, University of Jena
Organization: University of Jena (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GERMAIN; 2012-003023-38 (EudraCT Number)
Record Dates: First submitted 2013-08-13; First posted 2014-05-23 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Revlimid; Lenalidomide maintenance
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide 10mg/day
  Interventions: Drug: Lenalidomide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenalidomide — after 6 cycles VMP Patients will receive Lenalidomide given as two capsules 5 mg capsules p.o. daily until progressive disease (PD)
  Other Names: Revlimid
  Arms: Lenalidomide
Drug: Placebo — after 6 cycles VMP Patients will receive Placebo given as two capsules 5 mg capsules p.o. daily until progressive disease (PD)
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, blinded, 2-arm phase IIb trial that will compare the efficacy and safety of Lenalidomide maintenance after Bortezomib/Melphalan/Prednison (VMP) induction to VMP without maintenance (Placebo). In addition the trial will assess the treatment of Revlimid/low dose Dexamethasone (Rd) as Salvage after VMP without sufficient response (less than PR) in an observational arm. Key eligibility criteria include patients with newly diagnosed multiple myeloma and who are 65 years of age or older or are not candidates for high-dose chemotherapy and autologous stem cell transplantation. Patients with poor performance status or serious coexistent medical conditions will be excluded from this study. After registration all patients receive 6 cycles VMP (modified according to Mateos et al.). Patients who receive at least a PR and completed VMP can be randomized to either Lenalidomide 10 mg/d continuously maintenance or to placebo. Randomization will be stratified according to the quality of response after VMP induction (PR vs. VGPR + stringent complete remission [sCR] + CR). Patients that are not able to complete VMP due to toxicity but reached at least a PR after a minimum of four cycles of therapy should immediately proceed to randomization. Blinded phase continues until progression or end of study. After unblinding, patients who received placebo should be treated with Rd.

Patients that do not reach PR after induction with VMP or are progressive during treatment with VMP should not be randomized, but switched to the observation arm and treated with Rd immediately. The study treatment ends with the confirmed progression on maintenance treatment (Lenalidomide or placebo) for patients that reached PR with induction treatment, or with the confirmed progression on second-line therapy with Revlimid® and Dexamethasone for patients that did not reach PR on induction treatment. All patients will be followed up every 3 months after end of study treatment, until end of study. The study ends two years after Last Patient In (i.e. randomization for maintenance) if sufficient events for the primary endpoint were received, but not later than 8 years after trial initiation (whatever comes first).

DETAILED DESCRIPTION:
Primary objective

- Estimate the gain in progression-free survival (PFS) by maintenance with Lenalidomide after induction with VMP in elderly patients or patients unfit for highdose chemotherapy in comparison with placebo after VMP

Secondary study objectives

* To compare response rates of VMP and Lenalidomide maintenance versus VMP and placebo
* To compare overall survival probabilities between patients treated with Lenalidomide maintenance and patients without maintenance treatment
* To compare the safety of VMP and Lenalidomide maintenance versus VMP and placebo
* To compare the QoL of VMP and Lenalidomide maintenance versus VMP and placebo
* To assess the safety and efficacy of Rd for poor responders on VMP

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form.
2. Must be ≥18 years of age at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Previously untreated, symptomatic multiple myeloma as defined by the 3 criteria below:

   * Multiple Myeloma (MM) diagnostic criteria (all 3 required):

     * Monoclonal plasma cells in the bone marrow ≥10% and/or presence of a biopsy-proven plasmacytoma
     * Monoclonal protein present in the serum and/or urine
     * Myeloma-related organ dysfunction (at least one of the following):

       * [C] Calcium elevation in the blood (serum calcium >10.5 mg/dl or upper limit of normal)
       * [R] Renal insufficiency (serum creatinine >2 mg/dl)
       * [A] Anemia (hemoglobin <10 g/dl or 2 g < laboratory normal)
       * [B] Lytic bone lesions or osteoporosis

   AND have measurable disease by protein electrophoresis analyses as defined by the following:
   * Immunoglobulin (Ig)G multiple myeloma: Serum monoclonal paraprotein (M-protein) level
   * 1.0 g/dl or urine M-protein level - 200 mg/24 hours
   * IgA multiple myeloma: Serum M-protein level - 0.5 g/dl or urine Mprotein level - 200 mg/24 hours
   * IgM multiple myeloma (IgM M-protein plus lytic bone disease documented by skeletal survey plain films): Serum M-protein level ≥ 1.0 g/dl or urine M-protein level ≥ 200mg/24hours
   * IgD multiple myeloma: Serum M-protein level - 0.05 g/dl or urine Mprotein level - 200 mg/24 hours
   * Light chain multiple myeloma: Serum M-protein level - 1.0 g/dl or urine M-protein level - 200 mg/24 hours

   AND are at least 65 years of age or older or, if younger than 65 years of age, are not candidates for stem cell transplantation because:
   * The patient declines to undergo stem cell transplantation

   OR:
   * Stem cell transplantation is not available to the patient
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
6. Female of childbearing potential (FCBP) † must:

   * Understand the potential teratogenic risk to the unborn child
   * Understand the need for effective contraception, without interruption, 4 weeks before starting study treatment, throughout the entire duration of study treatment, dose interruption and 28 days after the end of study treatment
   * Be capable of complying with effective contraceptive measures and agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 28 days after study treatment discontinuation. The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. FCBP must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:

     * Highly effective methods*:

       * Intrauterine device (IUD)**
       * Progesterone only hormonal contraceptive (birth control pills, injections, implants)*
       * Tubal ligation
       * Partner's vasectomy
     * Additional effective methods:

       * Male condom (partner)
       * Diaphragm
       * Cervical Cap
   * (*)Because of the increased risk of venous thromboembolism in patients with multiple myeloma taking Lenalidomide and Dexamethasone, combined oral contraceptive pills are not recommended. If a patient is currently using combined oral contraception she should switch to one of the effective method listed above. The risk of venous thromboembolism continues for 4 to 6 weeks after discontinuing combined oral contraception. The efficacy of contraceptive steroids may be reduced during co-treatment with Dexamethasone.
   * (**)Implants and levonorgestrel-releasing intrauterine systems are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered particularly in patients with neutropenia.
   * Be informed about and understand the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy
   * Agree to have two medically supervised pregnancy tests with a minimum sensitivity of 25 mIU/ml (milli-International Units per milliliter) prior to starting Lenalidomide. The first pregnancy test must be performed within 10 to 14 days prior to the start Lenalidomide and the second pregnancy test must be performed within 24 hours prior to the start of Lenalidomide. The patient will receive Lenalidomide only after the study doctor has verified that the results of these pregnancy tests are negative. She must understand the need to commence the study treatment as soon as study drug is dispensed following the second negative pregnancy test. This requirement also applies to FCBP who practice complete and continued abstinence.
   * Must understand the need and accepts to undergo pregnancy testing in the frequency as follows: FCBP with regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at day 28 following study drug discontinuation. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following study drug discontinuation. This requirement also applies to FCBP who practice complete and continued abstinence.
   * Females must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation.

A FCBP † is a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months).

Male subjects must:

* Understand the potential teratogenic risk if engaged in sexual activity with a pregnant female or a FCBP
* Understand the need for the use of a condom and agree to use condoms even if he has had a vasectomy, if engaged in sexual activity with a pregnant female or a female of childbearing potential , while taking study drug, during any dose interruptions and for 28 days after stopping study therapy.
* Agree to notify the investigator immediately, if pregnancy or a positive pregnancy test occurs in his partner during study participation.
* Agree to abstain from donating semen or sperm during therapy or for at least 28 days following discontinuation of study drug.

All subjects must:

* Agree to abstain from donating blood while taking study drug therapy and for at least 28 days following discontinuation of study drug therapy.
* Agree never to give Lenalidomide to another person and to return all unused study drug to the investigator.

Exclusion Criteria:

1. Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid [i.e., less than or equal to the equivalent of Dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 14 days of registration]).
2. Any serious medical condition that places the patient at an unacceptable risk if he or she participates in this study. Examples of such a medical condition are, but are not limited to, patient with unstable cardiac disease as defined by: Cardiac events such as MI within the past 6 months, NYHA (New York Heart Association) heart failure class III-IV, uncontrolled atrial fibrillation or hypertension; patients with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis and lupus, that likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
3. Pregnant or breast feeding females.
4. Any of the following laboratory abnormalities within 1 week prior to registration:

   * Absolute neutrophil count (ANC) < 1,000/µL (1.0 x 109/L) without the use of colony stimulating factors within 14 days before the laboratory test. Untransfused platelet count < 50,000 cells/µL (50 x 109/L)
   * Hemoglobin < 7.5 g/dL (4.6 mmol/L) (regardless of transfusion support or prior medication with erythropoietin)
   * Serum sGOT/AST (serum glutamic-oxaloacetic transaminase/ aspartate aminotransferase) or SGPT(serum glutamate pyruvate transaminase)/ALT > 3.0 x upper limit of normal (ULN)
   * Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L)
5. Renal failure with creatinine clearance (CLCR)< 15 ml/min or requiring hemodialysis or peritoneal dialysis.
6. Psychiatric illness that would prevent the subject from signing the informed consent form or from completion of treatment according to the protocol.
7. Patient currently is enrolled in another clinical research study or has been enrolled in such a study within 4 weeks before randomization/registration and/or is receiving an investigational agent for any reason or has received such an agent within 4 weeks before registration.
8. Prior history of malignancies, other than multiple myeloma, unless the patient has been free of the disease for 3 years. Exceptions include the following, if treated with curative intent:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
9. Known positive for HIV or active hepatitis A, B or C viral infection.
10. Immunotherapy or antibody therapy within 8 weeks before registration.
11. Major surgery within 4 weeks before registration.
12. Any severe systemic infection requiring treatment.
13. Patients who are unable or unwilling to undergo antithrombotic therapy.
14. Peripheral neuropathy of ≥ grade 3 severity or grade 2 severity with pain.
15. Primary AL (amyloid light chain) amyloidosis and myeloma complicated by amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Median Progression free survival | maximum of 8 years
  time from randomization to the first documentation of disease progression or death due to any cause, whichever comes first, assessed up to the end of the study (maximum of 8 years)

SECONDARY OUTCOMES:
overall survival | 5 years after randomization
sequence progression-free survival | maximum of 8 years
  defined as time from initial registration before start of VMP treatment to the first documentation of disease progression based on the International Myeloma Working Group (IMWG) criteria, or death due to any cause during the study up to the end of the PFS follow-up phase
efficacy parameters according to the international uniform response criteria | after VMP (31 weeks) and 6 months of maintenance or placebo
  complete response [CR], stringent complete response [sCR], very good partial response (VGPR), partial response [PR], and overall response [CR + VGPR + PR] using IMWG criteria
number and indication of adverse events | maximum of 8 years
  time of first study treatment until up to the end of the follow-up phase (maximum of 8 years)
Quality of life | maximum of 8 years
  initial registration up to the end of the follow-up phase (maximum of 8 years), European Organization for Research and Treatment of Cancer (EORTC) QLQ (Quality of Life)-C30, QLQ-MY20 (Myeloma 20), EQ (European Questionnaire)-5D
Time to treatment failure | maximum 8 years
  defined as a composite endpoint measuring time from randomization to discontinuation of study treatment for any reason, including disease progression, treatment toxicity, start of another anti-myeloma treatment, and death, whichever comes first
sequence overall survival | maximum of 8 years
  time from registration before start of VMP treatment until death due to any cause or until censoring at the last time the patient was known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Brioli, MD, Principal Investigator — Jena University Hospital
Locations (19):
- Germany (19):
  - Charité - Campus Benjamin Franklin Medizinische Klinik II, Berlin
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Gemeinschaftspraxis Mohm / Prange-Krex, Dresden
  - Onkologische Schwerpunktpraxis, Dresden
  - Internistische Gemeinschaftspraxis, Güstrow
  - Universitätsklinkum Halle, Halle
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Abt. Hämatologie und internistische Onkologie, Jena
  - Universitätsklinikum Leipzig, Department für Innere Medizin, Leipzig
  - Dr. Aldaoud - Dr. Schwarzer Forschungsgesellschaft mbH, Leipzig
  - Gemeinschaftspraxis Uhle, Müller, Kröning, Jentsch-Ullrich, Magdeburg
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Universitätsmedizin Rostock, Rostock
  - Klinikum Südstadt Rostock, Rostock
  - Johanniter-Krankenhaus Gethin-Stendal GmbH, Stendal
  - Medizinisches Versorgungszentrum GmbH, Weiden
  - Universitätsklinikum Würzburg, Würzburg
  - Heinrich-Breun-Klinikum gGmbH, Zwickau

IPD SHARING:
Plan to Share IPD: No